CLINICAL TRIAL: NCT03398356
Title: The Assessment of the Effect of Metformin and Its Serum Concentration on the Concentration of Substances Associated With the Production of Nitric Oxide in Patients With Impaired Carbohydrate Metabolism
Brief Title: Metformin and Its Impact on the Substances Associated With NO Production in Prediabetes Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Edyta Sutkowska, MD, PhD; The Head of the Department and Division of Medical Rehabilitation, Wroclaw Medical University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ST.C310.17.009
Record Dates: First submitted 2018-01-07; First posted 2018-01-12 (Actual); Results first posted 2020-08-24 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: PreDiabetes; Impaired Fasting Glucose (IFG); Impaired Glucose Tolerance (IGT)
Keywords: prediabetes; impaired fasting glucose; impaired glucose tolerance; metformin; nitric oxide
MeSH Terms: conditions — Prediabetic State; Glucose Intolerance | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: The group of patients taking the drug at the target dose of 3 x 1000 after 4 weeks returned to the dose of 3 x 500 mg. The group of patients taking the drug at the target dose 3 x 500 mg consequently had this dose during the whole study period.
  The basic parameters and biochemical parameters from healthy individuals at the beginning of the study were assessed to compare with patients with pre-diabetes. This group did not take the metformin and thus did not have further examination and lab-tests during the study.
Who Masked: Investigator
Masking Description: At the beginning of the study, patients are assigned a number by a nurse and are assigned to group A or B according to ID. When analyzing the results, the researchers only knows the numbers of blood samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group A (Other): metformin dose 3 x 500 mg
  Interventions: Drug: Metformin
- group B (Other): metformin dose 3 x 1000 mg
  Interventions: Drug: Metformin
- group C (No Intervention): healthy volunteers who had basic parameters assessment and blood tests only at the beginning of the study

INTERVENTIONS:
Drug: Metformin — for group A: 12 weeks metformin treatment in a final dose 3 x 500 mg
  for group B: 3 weeks metformin treatment in a dose 3 x 500 mg, next: 3 weeks metformin treatment in a final dose 3 x 1000mg, next: 3 weeks metformin treatment in a dose 3 x 500 mg.
  Other Names: Metformax; Glucophage; Formetic; Siofor
  Arms: group A; group B

SUMMARY:
This study evaluates the effect of different doses of metformin on the function of endothelium in people with pre-diabetes. One group of the patients will receive metformin in dose: 1500 mg, the second one will receive 3000 mg/day.

The parameters from healthy volunteers will be taken only at the study beginning to compare the test results with the parameters from patients with pre-diabetes. This group will be not treated with metformin (no intervention)

DETAILED DESCRIPTION:
In addition to exercise and diet, metformin is a medicine used to treat diabetes mellitus (DM) and pre-diabetic (pre-DM) conditions. This drug improves insulin sensitivity in both groups of patients (DM and pre-DM) and as a result gives a reduction in blood glucose.

However, studies also confirm the effect of metformin on the reduction of cardiovascular risk in patients with diabetes (UKPDStudy), regardless of the hypoglycaemic effect.

The precise mechanism of action of the drug in this field is not clear. There is also no data on whether similar effects apply to patients with pre-diabetes. Although we know that this group of patients is also characterized by increased cardiovascular risk.

One of the most important substances that are involved in vasodilation is nitric oxide (NO). Impairment of its secretion is an important signal of endothelial damage and is connected with cardiovascular complications.

The impact of metformin on endothelial function in pre-diabetes patients is not known. We do not know the effect of the drug dose and its different serum concentration on the secretion of the dilators of the vessels, which are associated with endothelial function.

The study involves patients with pre-diabetes who meet the inclusion criteria, have no contraindication to participate in the study (see exclusion criteria), and give their written consent after reading "Information for the patient".

The conditions (IFG, IGT) for participation in the study are confirmed by a diabetologist (principal investigator ) based on fasting glucose and OGTT (oral glucose tolerance test) with 75 mg of glucose.

Metformin will be given in an increasing dose in accordance with the test protocol.

After reaching a one-week treatment with a dose of 3 x 500 mg, patients will be assigned to group A -a continuation of a dose of 3 x 500 and group B- increase dose to 3 x 1000mg. Randomization depends on the identification number (ID). The patients with an even, second number in the PESEL (identification number) will be randomized to the A group, the patients with the second, odd number in the PESEL will be randomized to the group B. Here as an example: PESEL: 60010102823-" 0" is as an even number so the patient will be randomized to the group A; PESEL: 61010102823- "1" is an odd number- the patient will be randomized to the group B. This PESEL number (ID) in Poland is given to every person shortly after birth and the researchers have no influence on it.

In the final stage also patients from group B (metformin: 3 x 1000 mg), will back to the treatment dose of metformin 3 x 500 mg- to show the relationship between the dose, serum concentration of the metformin and its effect on the secretion of the measured substances.

The healthy volunteers will be not treated with metformin. Patients will be reminded by phone about the increase in metformin dose as well as on control visits.

The lack of possible treatment with proper doses of metformin due to poor drug tolerance will move the patient from group B to group A if such dose (3 x 500 mg) is well tolerated. The patient will be excluded from the study if no compliance or lack of contact with the patient will be recorded during the treatment period or if metformin dose: 3 x 500 mg will be characterized with bad tolerance.

Information about: age, gender, BMI, cardiovascular risk factors, the current basic lab-tests, and pharmacotherapy will be recorded.

The blood samples for: plasma metformin level and listed substances will be collected for patients with pre-diabetes as described below (see diagram). The basic parameters as well as NO indirect products concentrations will be assessed for healthy volunteers only once-at the beginning of the study.

Test 1: NO(0) (indirect products) for patients before treatment start

3 weeks increasing dose of metformin to the final dose: 1500mg/day

3 x 500 mg (1500/day)- the dose is reached

3 weeks treatment 1500mg/day

Tests 2: NO1(1500) and metformin concentration

Randomization B:3 weeks increasing dose A: 6 weeks continuation with of metformin to the final a dose 3 x 500 mg

dose 3 x 1000mg

3 x 1000mg (3000mg/day)- the dose is reached 3 weeks treatment 3000mg/day Tests 3: NO2(1000) or NO3(500) and metformin concentration for both groups

3 weeks treatment 1500mg/day for both groups

Test 4: NO4 and metformin concentration

Statistical analysis:

For statistical analysis, the Statistica 12 program will be used (StatSoft Polska Sp. z o.o. www.statsoft.pl).

The cut-off point for statistical significance (p) was determined at 0.05. To determine the statistical significance will be used tests compliant with the distribution of variables and data character (Student's t-test, Mann-Whitney test, chi-square test, Kruskal-Wallis ANOVA test). For analysis taking into account the duration of the study and determine the impact of relevant variables to achieve the appropriate concentration of nitric oxide will be used Cox proportional hazard regression. The goal of the optimal determination cut-off point for predictors will use ROC curves. Logistic regression was used to determine the independent predictors to obtain the desired concentration of nitric oxide. In order to determine the correlation, it will be used correlation of order Spearman's rank correlation coefficient or Pearson correlation coefficient.

ELIGIBILITY:
Inclusion Criteria for treated groups ( A or B):

* age: 40-65 years;
* pre-diabetic status based on fasting plasma glucose (FPG) and / or OGTT;
* without metformin before;
* without ischemic heart disease in history;
* without a stroke in a history;
* without PAOD (peripheral arterial occlusive disease) in a history;
* without active cancer in a history

Exclusion Criteria for treated groups (A or B):

* age <40 or >65;
* diabetes;
* taking metformin before study;
* active cancer;
* history of macro-angiopathy (ischemic heart disease, stroke or TIA, PAOD);
* serious gastrointestinal disease that may affect metformin tolerance;
* renal failure with GFR<45 ml/min/1.73m2;
* alanin transaminase > 3 x ULN

Inclusion criteria for healthy volunteers:

* age: 40-65 years;
* no carbo-hydrates disturbances (based on fasting plasma glucose (FPG) and/or OGTT);
* without metformin before;
* without ischemic heart disease in history;
* without a stroke in a history;
* without PAOD (peripheral arterial occlusive disease) in a history;
* without active cancer in a history

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edyta Sutkowska, PhD, Principal Investigator — Wroclaw Medical University
Locations (1):
- NZOZ Nowy Dwór, Wroclaw, Lower Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary outcome will be made available.
Supporting Information: Study Protocol, SAP
Time Frame: the results will be available after the publication of the study
Access Criteria: data will be available after giving permission by the Investigator

REFERENCES:
- [Background] IDF Clinical Guidelines Task Force. Global Guideline for Type 2 Diabetes: recommendations for standard, comprehensive, and minimal care. Diabet Med. 2006 Jun;23(6):579-93. doi: 10.1111/j.1464-5491.2006.01918.x. PMID 16759299
- [Background] Nathan DM, Buse JB, Davidson MB, Heine RJ, Holman RR, Sherwin R, Zinman B; Professional Practice Committee, American Diabetes Association; European Association for the Study of Diabetes. Management of hyperglycaemia in type 2 diabetes: a consensus algorithm for the initiation and adjustment of therapy. A consensus statement from the American Diabetes Association and the European Association for the Study of Diabetes. Diabetologia. 2006 Aug;49(8):1711-21. doi: 10.1007/s00125-006-0316-2. No abstract available. PMID 16802130
- [Background] Effect of intensive blood-glucose control with metformin on complications in overweight patients with type 2 diabetes (UKPDS 34). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):854-65. PMID 9742977
- [Background] Hamed S, Brenner B, Roguin A. Nitric oxide: a key factor behind the dysfunctionality of endothelial progenitor cells in diabetes mellitus type-2. Cardiovasc Res. 2011 Jul 1;91(1):9-15. doi: 10.1093/cvr/cvq412. Epub 2010 Dec 24. PMID 21186243
- [Background] De Jager J, Kooy A, Lehert P, Bets D, Wulffele MG, Teerlink T, Scheffer PG, Schalkwijk CG, Donker AJ, Stehouwer CD. Effects of short-term treatment with metformin on markers of endothelial function and inflammatory activity in type 2 diabetes mellitus: a randomized, placebo-controlled trial. J Intern Med. 2005 Jan;257(1):100-9. doi: 10.1111/j.1365-2796.2004.01420.x. PMID 15606381
- [Background] Wisniewski J, Fleszar MG, Piechowicz J, Krzystek-Korpacka M, Chachaj A, Szuba A, Lorenc-Kukula K, Maslowski L, Witkiewicz W, Gamian A. A novel mass spectrometry-based method for simultaneous determination of asymmetric and symmetric dimethylarginine, l-arginine and l-citrulline optimized for LC-MS-TOF and LC-MS/MS. Biomed Chromatogr. 2017 Nov;31(11). doi: 10.1002/bmc.3994. Epub 2017 May 24. PMID 28436051
- [Result] Sutkowska E, Fortuna P, Wisniewski J, Sutkowska K, Hodurek P, Gamian A, Kaluza B. Low metformin dose and its therapeutic serum concentration in prediabetes. Sci Rep. 2021 Jun 3;11(1):11684. doi: 10.1038/s41598-021-91174-7. PMID 34083618
- [Result] Sutkowska E, Fortuna P, Kaluza B, Sutkowska K, Wisniewski J, Prof AG. Metformin has no impact on nitric oxide production in patients with pre-diabetes. Biomed Pharmacother. 2021 Aug;140:111773. doi: 10.1016/j.biopha.2021.111773. Epub 2021 May 29. PMID 34062418
- [Result] Sutkowska E, Fortuna P, Kaluza B, Sutkowska K, Hodurek P, Fleszar MG. The impact of Sample Handling Time on metformin serum concentration. Biomed Pharmacother. 2021 Jan;133:110971. doi: 10.1016/j.biopha.2020.110971. Epub 2020 Nov 25. PMID 33248407

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: metformin dose 3 x 500 mg
  Metformin: for group A: 12 weeks metformin treatment in a final dose 3 x 500 mg
  for group B: 3 weeks metformin treatment in a dose 3 x 500 mg, next: 3 weeks metformin treatment in a final dose 3 x 1000mg, next: 3 weeks metformin treatment in a dose 3 x 500 mg.
- Group B: metformin dose 3 x 1000 mg
  Metformin: for group A: 12 weeks metformin treatment in a final dose 3 x 500 mg
  for group B: 3 weeks metformin treatment in a dose 3 x 500 mg, next: 3 weeks metformin treatment in a final dose 3 x 1000mg, next: 3 weeks metformin treatment in a dose 3 x 500 mg.
- Group C: control healthy volunteers, no intervention
Period: Before Treatment
Arm/Group | Group A | Group B | Group C
Started | 15 | 21 | 11
Completed | 12 | 13 | 0 (only baseline parameters were taken, this group did not participate in the further part of the study)
Not Completed | 3 | 8 | 11
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — drug intolerance | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 5 | 0
Not completed — Physician Decision | 0 | 0 | 11
Period: After 6 Weeks of Treatment
Arm/Group | Group A | Group B | Group C
Started | 12 | 13 | 0 (control group- only initial parameters were assessed to compare, no follow-up)
Completed | 12 | 11 | 0 (control group- only initial parameters were assessed to compare, no follow-up)
Not Completed | 0 | 2 | 0
Not completed — Physician Decision | 0 | 2 | 0
Period: Post 6 Week Period Initial Evaluation
Arm/Group | Group A | Group B | Group C
Started | 14 (two of the patients were moved from group B, because of intolerance of the higher dose of the drug) | 11 | 0
Completed | 14 | 11 | 0
Not Completed | 0 | 0 | 0
Period: After 12 Weeks of Treatment
Arm/Group | Group A | Group B | Group C
Started | 14 | 11 | 0 (control group- only initial parameters were assessed to compare, no follow-up)
Completed (two of the patients were moved from group B, because of intolerance of the higher dose of the drug) | 14 | 11 | 0 (control group- only initial parameters were assessed to compare, no follow-up)
Not Completed | 0 | 0 | 0
Period: After 15 Weeks of Treatment
Arm/Group | Group A | Group B | Group C
Started | 14 | 11 | 0 (control group- only initial parameters were assessed to compare, no follow-up)
Completed | 14 | 11 | 0 (control group- only initial parameters were assessed to compare, no follow-up)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: group C was a comparator only for baseline parameters
Groups:
- Group A: Patients with pre-diabetes; metformin dose 3 x 500 mg
  Metformin: for group A: 12 weeks metformin treatment with a final dose 3 x 500 mg, after 3 weeks of the titration Total treatment time: 15 weeks
- Group B: Patients with pre-diabetes, max metformin dose 3 x 1000 mg
  Metformin: for group B: 3 weeks metformin treatment with a dose 3 x 500 mg, after 3 weeks of the titration next: 3 weeks metformin treatment with a final dose 3 x 1000mg, after 3 weeks of the titration next: 3 weeks metformin treatment with a dose 3 x 500 mg. Total treatment time: 15 weeks
- Group C: healthy volunteers
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 14 | 11 | 11 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.64 (8.85) | 55.73 (8.27) | 49.90 (8.37) | 51.97 (8.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 6 | 14
  Male | 9 | 8 | 5 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Poland | 14 | 11 | 11 | 36
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.49 (5.26) | 30.75 (4) | 26.99 (5.43) | 29.89 (5.21)
body mass [Mean (Standard Deviation); unit: kg] | 96.71 (13.74) | 92.36 (9.73) | 80.81 (20.64) | 90.52 (16.28)
creatinine [Mean (Standard Deviation); unit: mg/dl] | 0.86 (0.18) | 0.89 (0.16) | 0.73 (0.03) | 0.85 (0.16)
alanin transaminase [Mean (Standard Deviation); unit: U/l] | 28.13 (14.01) | 35.45 (20.51) | 19.11 (12.06) | 28.11 (16.74)
TCL- total cholesterol level [Mean (Standard Deviation); unit: mg/dl] | 207.21 (50.22) | 184.91 (34.19) | 201 (27.47) | 198.50 (39.71)
TG-triglicerydes [Mean (Standard Deviation); unit: mg/dl] | 133.29 (62.77) | 136.82 (66.63) | 137.09 (49.20) | 135.53 (58.54)
HDL- high density lipoprotein [Mean (Standard Deviation); unit: mg/dl] | 49.86 (12.07) | 50.73 (14.35) | 57.91 (16.82) | 52.58 (14.38)
LDL-low density lipoprotein [Mean (Standard Deviation); unit: mg/dl] | 125.29 (30.79) | 106.95 (23.78) | 115.70 (19.91) | 116.75 (26.20)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dl] | 109.39 (11.13) | 107.23 (5.95) | 88.81 (4.44) | 102.44 (12.11)
liver steatosis [Count of Participants; unit: Participants] — assessed by ultrasonography as Yes or No
  Participants | 7 | 9 | 1 | 17
nicotinism [Count of Participants; unit: Participants] — active smoker- based on the patient's relation: Yes or No
  Participants | 3 | 4 | 2 | 9
hypertension [Count of Participants; unit: Participants] — based on patient's relation or information from the medical-records
  Participants | 7 | 6 | 3 | 16
family history for DM [Count of Participants; unit: Participants] — based on the patient's relation: first-line relatives: Yes or No
  Participants | 7 | 4 | 3 | 14
arginine [Mean (Standard Deviation); unit: µM] — LC-MS/MS (liquid chromatography-mass spectrometry) technique
  µM | 114.29 (28.15) | 110.37 (27.63) | 122.11 (27.96) | 115.48 (27.54)
ADMA [Mean (Standard Deviation); unit: µM] — LC-MS/MS (liquid chromatography-mass spectrometry) technique
  µM | 0.51 (0.09) | 0.53 (0.09) | 0.56 (0.10) | 0.53 (0.09)
SDMA [Mean (Standard Deviation); unit: µM] — LC-MS/MS (liquid chromatography-mass spectrometry) technique
  µM | 0.39 (0.07) | 0.41 (0.10) | 0.42 (0.08) | 0.41 (0.08)
DMA [Mean (Standard Deviation); unit: µM] — LC-MS/MS (liquid chromatography-mass spectrometry) technique
  µM | 1.77 (0.71) | 1.74 (0.48) | 1.67 (0.40) | 1.73 (0.55)
Citrulline [Mean (Standard Deviation); unit: µM] — LC-MS/MS (liquid chromatography-mass spectrometry) technique
  µM | 34.10 (9.84) | 38.33 (7.49) | 36.45 (8.82) | 36.11 (8.8)
Ornithine [Mean (Standard Deviation); unit: µM] — LC-MS/MS (liquid chromatography-mass spectrometry) technique
  µM | 34.77 (11.58) | 37.12 (15.71) | 35.57 (11.09) | 35.73 (12.51)

OUTCOME MEASURES:

1. Primary Outcome: Serum Levels of Metformin at Different Time Points
Description: the serum concentration of the studied drug-metformin
Time Frame: 6 weeks from treatment start; 12 weeks from treatment start; 15 weeks from treatment start
Population: Group A and B- patients with pre-diabetes treated with different metformin dose (according to the information above as arm description) , group C- healthy volunteers, no metformin assessment as no treatment
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 14 | 11 | 0
µM
  6 weeks from the start of treatment | 4.36 (2.36) | 4.25 (2.58) |
  12 weeks from the start of treatment | 5.09 (2.29) | 7.42 (4.77) |
  15 weeks from the start of treatment | 4.66 (3.73) | 4.01 (4.01) |

2. Primary Outcome: Serum Levels of Arginine at Different Time Points
Description: arginine serum concentration
Time Frame: Baseline; 6 weeks from treatment start; 12 weeks from treatment start; 15 weeks from treatment start
Population: Groups A and B -patients with pre-diabetes treated with different dose of the metformin, group C- healthy volunteers, no metformin
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 14 | 11 | 0
µM
  6 weeks from the start of treatment | 112.18 (53.42) | 111.72 (36.89) |
  12 weeks from the start of treatment | 107.72 (13.93) | 97.69 (38.76) |
  15 weeks from the start of treatment | 104.72 (34.21) | 103.76 (19.76) |

3. Primary Outcome: Serum Levels of ADMA at Different Time Points
Description: ADMA- asymmetric dimethylarginine-serum concentration
Time Frame: before study start; 6 weeks from treatment start; 12 weeks from treatment start; 15 weeks from treatment start
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 14 | 11 | 0
µM
  6 weeks from the start of treatment | 0.51 (0.11) | 0.57 (0.11) |
  12 weeks from the start of treatment | 0.52 (0.09) | 0.55 (0.14) |
  15 weeks from the start of treatment | 0.50 (0.08) | 0.52 (0.10) |

4. Primary Outcome: Serum Levels of SDMA at Different Time Points
Description: SDMA-symmetric dimethylarginine-serum concentration
Time Frame: Baseline; 6 weeks from treatment start; 12 weeks from treatment start; 15 weeks from treatment start
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 14 | 11 | 0
µM
  6 weeks from the start of treatment | 0.40 (0.08) | 0.45 (0.08) |
  12 weeks from the start of treatment | 0.41 (0.08) | 0.42 (0.08) |
  15 weeks from the start of treatment | 0.39 (0.07) | 0.39 (0.06) |

5. Primary Outcome: Serum Levels of Citrulline at Different Time Points
Description: serum concentration of the citrulline
Time Frame: Baseline; 6 weeks from treatment start; 12 weeks from treatment start; 15 weeks from treatment start
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 14 | 11 | 0
µM
  6 weeks from the start of treatment | 21.73 (6.66) | 28.08 (11.31) |
  12 weeks from the start of treatment | 25.95 (9.48) | 27.01 (15.38) |
  15 weeks from the start of treatment | 26.93 (9.71) | 29.77 (11.26) |

6. Primary Outcome: Serum Levels of DMA at Different Time Points
Description: DMA- dimethylamine, serum concentration
Time Frame: Baseline; 6 weeks from treatment start; 12 weeks from treatment start; 15 weeks from treatment start
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: µM
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 14 | 11 | 0
µM
  6 weeks from the start of treatment | 1.71 (0.31) | 2.07 (0.52) |
  12 weeks from the start of treatment | 1.63 (0.28) | 1.89 (0.43) |
  15 weeks from the start of treatment | 1.62 (0.34) | 1.84 (0.68) |

ADVERSE EVENTS:
Time Frame: 15 weeks
Description: Other- important gastrointestinal side effects which did not allow the prescribed dose to be continued
Groups:
- Group C: healthy volunteers, no intervention
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/21 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/21 | 0/11
Other Adverse Events (participants affected / at risk) | 3/15 | 2/21 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=15) | Group B (N=21) | Group C (N=11)
drug intolerance (Gastrointestinal disorders) | 3 (3) | 2 (2) | NA — the side effect which did not allow the prescribed dose to be continued

LIMITATIONS AND CAVEATS:
We didn't differentiate pts according to sex or gender. Before the study was finished we assessed the correlation between metformin concentration and BMI/ body mass. It was prepared as an additional analysis based on 20 cases (not published yet).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-06-13): https://cdn.clinicaltrials.gov/large-docs/56/NCT03398356/Prot_SAP_ICF_000.pdf